CLINICAL TRIAL: NCT05704764
Title: IRIS: Intervention to Reduce Internalized Stigma (IRIS) Among People Living With HIV Who Use Substances
Brief Title: Using the Ending Self-Stigma Intervention to Reduce Internalized Stigma Among People Living With HIV Who Use Substances
Acronym: IRIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: University of Maryland (Other); National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRIS-ESS-HSU; R34DA055532 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-03

CONDITIONS: HIV; Stigma, Social; Substance Use
Keywords: cognitive behavioral therapy; social cognitive theory; stigma
MeSH Terms: conditions — Social Stigma; Substance-Related Disorders | interventions — Seroconversion

STUDY DESIGN:
Intervention Model Description: Two group randomized (1:1) design contrasting minimally enhanced treatment-as-usual (ME-TAU) with the IRIS intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Enhanced TAU (No Intervention): Participants assigned to the minimally enhanced treatment-as-usual condition will receive an educational pamphlet about internalized stigma to read at their leisure and will be encouraged to continue in all their customary HIV- and substance use-related services.
- IRIS (Experimental): Using the materials developed during study phase one, five approximately 60-90 minute sessions will be carried out with the 35 participants randomized to receive IRIS. Each by session will be administered by a trained interventionist and will be carried out over a virtual platform (e.g., Zoom, Teams). The sessions are based on cognitive behavioral therapy and social cognitive theory, and are intended to reduce negative thoughts about the self and improve self-efficacy to engage with HIV and substance use treatment. Any session hand-outs will be mailed and/or emailed to participants prior to each session and shared onscreen. Participants in the IRIS condition may also receive study-provided journals to supplement their IRIS experience.
  Interventions: Behavioral: Ending Self Stigma for Persons living with HIV and Use Substances

INTERVENTIONS:
Behavioral: Ending Self Stigma for Persons living with HIV and Use Substances — One-on-one intervention based on principles of cognitive behavioral therapy and social cognitive theory designed to reduce internalized stigma related to HIV and/or drug use.
  Other Names: IRIS
  Arms: IRIS

SUMMARY:
The goal of this clinical trial is to test an intervention to reduce stigma among people living with HIV who use opioids and cocaine. The main question it aims to answer is:

- Does reducing internalized stigma about HIV and/or drug use lead to improved HIV care outcomes?

After a year spent adapting an existing intervention to be applied specifically among people living with HIV who use substances, 70 participants will be randomized to receive either treatment-as-usual or the newly adapted intervention. The intervention itself will consist of five one-on-one sessions with a trained interventionist to discuss and work through the stigmas people commonly associate with HIV and/or substance use.

DETAILED DESCRIPTION:
Different types of stigma (e.g., anticipated, enacted, internalized) associated with illicit substance use (SU) and HIV positive status impede HIV treatment outcomes (incl. HIV healthcare retention, antiretroviral therapy [ART] adherence and viral load suppression). The premise of this study is that individuals can learn to diminish the personal effects of public stigma, thereby reducing internalized stigma and improving expected health outcomes.

To this end, this study adapted an existing evidence-based stigma reduction intervention, Ending Self-Stigma (ESS), which has shown efficacy in reducing internalized and anticipated stigma in populations experiencing mental health challenges, to be applied specifically among people living with HIV and using drugs and/or alcohol (or are currently in treatment for substance use). The new one-on-one intervention is IRIS, and it uses cognitive behavioral therapy strategies and social cognitive theory constructs to facilitate reductions in internalized stigma.

In the first phase, an iterative process beginning with formative interviews with service delivery key informants and people living with HIV/AIDS (PLWH) who use substances generated an initial version of IRIS. Intervention content was adapted based on participant feedback and intervention delivery was adapted for a virtual format.

In the second phase, a small pilot of the newly created IRIS intervention was carried out with persons living with HIV and using substances. Feedback from participants and intervention staff were used to refine the IRIS intervention.

In the third phase, a clinical trial testing the newly adapted IRIS intervention will be carried out with 70 participants (Group 1: Minimally Enhanced Treatment-as-Usual; Group 2: IRIS; 1:1 randomization) to determine feasibility and acceptability of the intervention in addition to collecting data on intervening variables (incl. internalized and anticipated stigma, depressive symptoms, anxiety, etc.).

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* English speaking
* Living with HIV
* Self-report recent drug and/or alcohol use OR currently enrolled in substance use treatment
* Willing and able to provide full informed consent
* Responds affirmatively to having ever experienced one or more of the following types of stigma related to HIV status or SU: (1) enacted, (2) anticipated, and/or internalized.

Exclusion Criteria:

* Does not meet all inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HIV-Related Internalized Stigma | 30 Days
  Change in Berger HIV Stigma scale scores (1 to 4, with higher scores meaning more internalized stigma)
Substance Use-Related Internalized Stigma | 30 days
  Changes in Substance Use Stigma Mechanism scores (1 to 5, with higher scores meaning more internalized stigma)

SECONDARY OUTCOMES:
ART Adherence | 30 days
  Change in self-reported ART adherence (5-point scale, with larger numbers meaning better ART adherence)
Mental Health Symptoms | 7 days
  Changes in CES-D (1 to 4, with larger numbers meaning more depression symptoms) and Spielberger Anxiety (1 to 4, with larger numbers meaning more anxiety) scale scores.
Intervention Satisfaction | 30 days
  Participant intervention satisfaction scores (1 to 5, with larger numbers meaning greater intervention satisfaction)
Substance Use | 30 days
  Self-reported days of substance use

CONTACTS AND LOCATIONS:
Overall Officials: Jesse B Fletcher, Ph.D., Principal Investigator — Friends Research Institute, Inc.; Alicia Lucksted, Ph.D., Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - Friends Research Institute, Inc. Satellite Office, Newhall, California
  - University of Maryland School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided